CLINICAL TRIAL: NCT00982280
Title: An Evaluation of the Effectiveness and Tolerability of Tapentadol Hydrochloride Prolonged Release, and Tapentadol Hydrochloride Immediate Release on Demand, in Subjects With Severe Chronic Pain Due to Osteoarthritis of the Knee Taking WHO Step III Analgesics But Showing a Lack of Tolerability.
Brief Title: Evaluation of Effectiveness and Tolerability of Tapentadol Hydrochloride in Subjects With Severe Pain Due to Osteoarthritis Taking WHO Step III Analgesics But Showing a Lack of Tolerability.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow Recruitment and supply of Investigational Medicinal Product Issues
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 847022; 2009-010425-39 (EudraCT Number)
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Results first posted 2011-12-14 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Chronic Pain; Osteoarthritis
Keywords: Osteoarthritis; pain assessment; tapentadol; centrally acting analgesic
MeSH Terms: conditions — Chronic Pain; Osteoarthritis | interventions — Tapentadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tapentadol (Experimental): Tapentadol PR was given orally twice a day. A maximum of 2 oral Tapentadol IR tablets per day, with a minimum of a 4 hour interval between doses, were taken if there were acute pain episodes. The total daily dose of Tapentadol PR and IR were not permitted to exceed 500 mg per day.
  Interventions: Drug: Tapentadol PR

INTERVENTIONS:
Drug: Tapentadol PR — Tapentadol Prolonged Release (PR) Titration and Optimal Dose Period: Starting at 50 mg, 100 mg or 150 mg Tapentadol PR twice daily, adjusting at 50 mg PR steps (upwards or downwards) as necessary to achieve a balance between pain relief and a satisfactory level of tolerability. Participants were not permitted to exceed 500 mg of Tapentadol per day.
  Maintenance Period: Participants continuing on the dose established in the previous period.
  Other Names: Nucynta; Palexia

SUMMARY:
The main objective of the study is to evaluate the effectiveness, tolerability, and safety of tapentadol hydrochloride prolonged release (PR) in participants suffering from severe chronic pain due to osteoarthritis of the knee who are taking WHO Step III analgesics and show lack of tolerability. This is a clinical effectiveness trial designed to establish a link between anticipated clinical outcomes and the clinical practice by means of selected measures of clinical and subject-reported outcome. The trial will compare the effectiveness of previous analgesic treatment (WHO Step III) with that of tapentadol hydrochloride PR treatment during defined periods of evaluation.

DETAILED DESCRIPTION:
The trial will last up to 13 weeks for each subject and includes:

* One week of observation under previous analgesic treatment.
* Twelve weeks of treatment with tapentadol hydrochloride PR.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have signed an Informed Consent Form indicating that they understand the purpose of and procedures required for the trial and are willing to participate in it.
* Participants are men or non-pregnant, non-lactating women. Sexually active women must be postmenopausal, surgically sterile, or practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double barrier method, contraceptive patch, male partner sterilization) before entry and throughout the trial. Women of childbearing potential must have a negative pregnancy test at screening.
* Participants must be appropriately communicative to verbalize and to differentiate with regard to location and intensity of the pain.
* Participants must be at least 40 years of age.
* Participants must have a diagnosis of osteoarthritis of the knee based on the American College of Rheumatology (ACR) Classification criteria:

  * Knee pain and
  * Radiographic osteophytes or
  * Knee pain and aged 40 years or above and
  * Morning stiffness of less than 30 minutes of duration and
  * Crepitus on motion.
* Participants must have pain at the reference joint which has been present for at least 3 months.
* Participant's pain must require a strong analgesic (defined as WHO Step III) as judged by the Investigator
* Participant must be taking a WHO Step III analgesic on a daily basis for at least 2 weeks prior to the Screening Visit.
* Participant must have responded to the WHO Step III analgesic, i.e., participant must have a confirmed average pain intensity score (NRS 3) of smaller or equal to 5 points during the last 3 days prior to the Screening Visit.
* Participant must report opioid-related side effects as the reason to change their analgesic
* Participant must report a rate of satisfaction with their previous analgesic regimen not exceeding "fair" on a subject satisfaction with treatment scale (5-point VRS).

Exclusion Criteria:

* Presence of a clinically significant disease or laboratory findings that in the Investigator's opinion may affect efficacy or safety assessments.
* Presence of active systemic or local infection that may, in the opinion of the Investigator, affect the efficacy, quality of life/function or safety assessments.
* History of alcohol or drug abuse, or suspicion thereof in Investigator's judgement.
* Presence of concomitant autoimmune inflammatory conditions.
* Known history of or laboratory values reflecting severe renal impairment.
* Known history of moderately or severely impaired hepatic function.
* History of or active hepatitis B or C within the past 3 months or history of HIV infection.
* History of seizure disorder or epilepsy.
* Any of the following within 1 year: mild/moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm. Severe traumatic brain injury within 15 years (consisting of 1 or more of the following: brain contusion, intracranial hematoma, either unconsciousness or post traumatic amnesia lasting more than 24 h) or residual sequelae suggesting transient changes in consciousness.
* Pregnant or breast-feeding.
* History of allergy to, or hypersensitivity to tapentadol hydrochloride or its excipients, or contraindications related to tapentadol hydrochloride including:
* participants with acute or severe bronchial asthma or hypercapnia.
* participants who have or are suspected of having paralytic ileus.
* Employees of the Investigator or trial site, with direct involvement in this trial or other trials under the direction of the Investigator or trial site, as well as family members of employees of the Investigator.
* Participation in another trial concurrently or within 4 weeks prior to the Screening Visit.
* Known to or suspected of not being able to comply with the protocol and the use of the investigational medicinal product.
* Use of monoamine oxidase inhibitors within 14 days before the Screening Visit.
* Non-stable dosing of selective serotonin reuptake inhibitors within 30 days before the Screening Visit (the doses must remain stable during the trial).
* Osteoarthritis in a flare state.
* Use of intra-articular injections of hyaluronic acid in the reference joint within 3 months before the Screening Visit.
* Presence of conditions other than OA of the reference joint that could confound the assessment or self-evaluation of pain, e.g., anatomical deformities, significant skin conditions such as abscess or syndromes with widespread pain such as fibromyalgia. Subjects with OA at joints other than the reference joint will not be excluded as long as the reference joint is the source of main pain and disability.
* History and clinical signs at the reference joint of crystal-induced (e.g., gout, pseudo-gout), metabolic, infectious and autoimmune disease.
* Any painful procedures during the trial (e.g., major surgery including the reference joint) that may, in the opinion of the Investigator, affect the efficacy or safety assessments.
* Pending litigation due to chronic pain or disability.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Hoggart, Dr. MD, Principal Investigator — FRCA, FRCAPM Heart of England NHS Trust
Locations (24):
- Australia (2):
  - Site 4, Melbourne
  - Site 2, Perth
- Denmark (5):
  - Site 4, Aalborg
  - Site 7, Hvidovre
  - Site 6, Kolding
  - Site 2, Odense
  - Site 3, Vejle
- Germany (5):
  - Site 1, Berlin
  - Site 7, Katzhütte
  - Site 2, Leer
  - Site 8, Leipzig
  - Site 9, Zerbst
- Poland (3):
  - Site 4, Lublin
  - Site 5, Ostrów Mazowiecka
  - Site 2, Tychy
- Spain (2):
  - Site 4, Madrid
  - Site 1, Valencia
- United Kingdom (7):
  - Site 3, Birmingham
  - Site 6, Carmarthen
  - Site 1, Leeds
  - Site 2, London
  - Site 8, Middlesbrough
  - Site 9, Oxford
  - Site 10, York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment of the first participant was on the 02 October 2009 and was prematurely terminated, due to slow recruitment, on 12 August 2010 (when the last subject completed the last follow-up examination).
Pre-assignment Details: The Trial had a duration of 13 weeks. The one week Observation Period did not involve dosing with Tapentadol. For Tapentadol analyses purposes the first 6 weeks of dosing with Tapentadol are reported as one period, Titration and Optimal Dose Period. The last 6 weeks on Tapentadol are reported as the Maintenance Period.
Groups:
- Tapentadol PR: All participants started with either 50 mg, 100 mg or 150 mg tapentadol hydrochloride PR (twice daily). The dose of tapentadol hydrochloride PR was adjusted to a level that provided adequate analgesia (upwards or downwards on a weekly basis as needed). After 5 weeks the doses of tapentadol hydrochloride PR was kept stable. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). Tapentadol hydrochloride IR 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes however, participants were not permitted to dose tapentadol hydrochloride IR once 500 mg tapentadol hydrochloride PR dose was reached.
Period: Observation Period
Arm/Group | Tapentadol PR
Started | 82
Completed | 63
Not Completed | 19
Not completed — Not eligible to be dosed | 19
Period: Titration and Optimal Dose Period
Arm/Group | Tapentadol PR
Started | 63
Completed | 55
Not Completed | 8
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 1
Period: Maintenance Period
Arm/Group | Tapentadol PR
Started | 55
Completed | 54
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 26
Region of Enrollment [Number; unit: participants]
  Spain | 4
  Poland | 16
  Denmark | 6
  Australia | 2
  Germany | 34
  United Kingdom | 1

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate
Description: Participants were considered responders if they reported the same or less average pain intensity over a 3 day period after 6 weeks of tapentadol PR treatment as with their previous analgesic treatment.
Time Frame: 6 weeks
Population: Per Protocol Set. Last Observation Carried Forward (LOCF).
Measure: Number; unit: Participants
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 53
Participants | 50

2. Secondary Outcome: Average Pain Intensity Before the Start of Tapentadol Treatment
Description: For this pain assessment, the participant was to indicate the level of average pain experienced over the previous 3 days on an 11-point Numerical Rating Scale(NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Baseline
Population: Intention to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 62
units on a scale | 4.7 (0.66)

3. Secondary Outcome: Change in Average Pain Intensity After 6 Weeks of Tapentadol PR Treatment.
Description: For this pain assessment, the participant was to indicate the level of average pain experienced over the previous 3 days on an 11-point Numerical Rating Scale(NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The value indicates the change from the baseline value on the 0 to 10 scale. A Negative value indicates a reduction in pain intensity from the baseline average pain intensity.
Time Frame: Baseline; Week 6 (6 weeks)
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 55
Units on a scale | -2.2 (1.55)

4. Secondary Outcome: Change in Average Pain Intensity After 12 Weeks of Tapentadol PR Treatment.
Description: as for outcome 3
Time Frame: Baseline; Week 12 (12 weeks)
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 32
Units on a scale | -2.7 (1.26)

5. Secondary Outcome: Baseline Western Ontario McMaster Questionnaire (WOMAC) Global Score Assessing Pain, Disability and Joint Stiffness of the Knee
Description: Western Ontario McMaster Questionnaire (WOMAC) Global Score: WOMAC is measured with a Likert ordinal scale (the participant gives one of 5 possible answers) A higher score indicate that a symptom is bothersome or disabling. The WOMAC is a self-administered questionnaire and has 24 questions: Pain, Stiffness and Physical Function. The possible scores range from 0-20 for pain, 0-8 for stiffness, 0-68 for physical function and these are then summed 0-96 for the global score. A lower score indicates a lower level of symptoms and or disability.
Time Frame: Baseline
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 62
Units on a scale | 54.2 (13.19)

6. Secondary Outcome: Change From Baseline in the Western Ontario McMaster Questionnaire (WOMAC) Global Score Assessing Pain, Disability and Joint Stiffness of the Knee Over the Last Week at Week 6
Description: The WOMAC is a self-administered questionnaire and has 24 questions: Pain, Stiffness and Physical Function. The possible scores range from 0-20 for pain, 0-8 for stiffness, 0-68 for physical function and these are then summed 0-96 for the global score. The negative value indicates that there has been an improvement since baseline, the higher the value the greater the change since baseline.
Time Frame: 6 weeks
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 55
Units on a scale | -24.5 (18.40)

7. Secondary Outcome: Change From Baseline in the Western Ontario McMaster Questionnaire (WOMAC) Global Score Assessing Pain, Disability and Joint Stiffness of the Knee Over the Last Week at Week 12
Description: as for outcome 6
Time Frame: 12 weeks
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 32
Units on a scale | -25.1 (16.10)

8. Secondary Outcome: EuroQol-5 (EQ-5D) Health Status Index Outcome Over Time
Description: The participant scored the EuroQol-5. This is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "full health" and 0 representing dead. The positive values indicate that during the study the health status improved.
Time Frame: 6 weeks
Population: Intention to treat (ITT).
Measure: Median (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 55
Units on a scale | 0.201 (0.288)

9. Secondary Outcome: EuroQol-5 (EQ-5D) Health Status Index Outcome Over Time
Description: as for outcome 8
Time Frame: 12 weeks
Population: Intention to treat (ITT).
Measure: Median (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 32
Units on a scale | 0.155 (0.291)

10. Secondary Outcome: Change in Health Related Quality of Life: EuroQol-5D Health State Visual Analog Scale (VAS)
Description: EuroQoL-5D Health State Visual Analog Scale (VAS) is a participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state. The values indicated represent the change from the baseline, a positive value indicates an improvement.
Time Frame: 6 Weeks
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 55
Units on a scale | 29.6 (15.3)

11. Secondary Outcome: Change in Health Related Quality of Life: EuroQol-5D Health State Visual Analog Scale (VAS)
Description: as for outcome 10
Time Frame: 12 Weeks
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 32
Units on a scale | 34.6 (17.9)

12. Secondary Outcome: Clinical Global Impression of Change
Description: In the Clinical Global Impression of Change (CGIC) the clinician indicates the perceived change over the treatment period. The clinician is requested to choose one of seven categories. Scores range from very much improved to very much worse.
Time Frame: Baseline; End of Week 6 (6 Weeks)
Population: Intention to treat (ITT).
Measure: Number; unit: participants
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 55
participants
  Very much improved | 6
  Much improved | 28
  Minimally improved | 18
  No change | 1
  Minimally worse | 2
  Much worse | 0
  Very much worse | 0

13. Secondary Outcome: Clinical Global Impression of Change
Description: as for outcome 12
Time Frame: Baseline; End of Week 12 (12 Weeks)
Population: Intention to treat (ITT).
Measure: Number; unit: participants
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 32
participants
  Very much improved | 3
  Much improved | 17
  Minimally improved | 11
  No change | 1
  Minimally worse | 0
  Much worse | 0
  Very much worse | 0

14. Secondary Outcome: Patient Global Impression of Change
Description: In the Patient Global Impression of Change (PGIC) the participant indicates the perceived change over the treatment period. The participant is requested to choose one of seven categories. Scores range from very much improved to very much worse.
Time Frame: Baseline; End of Week 6 (6 Weeks)
Population: Intention to treat (ITT).
Measure: Number; unit: participants
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 55
participants
  Very much improved | 6
  Much improved | 28
  Minimally improved | 18
  No change | 1
  Minimally worse | 2
  Much worse | 0
  Very much worse | 0

15. Secondary Outcome: Patient Global Impression of Change
Description: as for outcome 14
Time Frame: Baseline; End of Week 12 (12 Weeks)
Population: Intention to treat (ITT).
Measure: Number; unit: participants
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 32
participants
  Very much improved | 3
  Much improved | 17
  Minimally improved | 11
  No change | 1
  Minimally worse | 0
  Much worse | 0
  Very much worse | 0

16. Secondary Outcome: Participant's Satisfaction With Previous Analgesic Treatment.
Description: Participants were requested to rate their previous analgesic medication on a 5-point scale. Previous medication was rated as excellent, very good, good, fair and poor.
Time Frame: Baseline
Population: Intention to treat (ITT).
Measure: Number; unit: participants
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 62
participants
  Excellent | 0
  Very Good | 0
  Good | 1
  Fair | 46
  Poor | 15

17. Secondary Outcome: Participant's Satisfaction With New Analgesic Treatment, i.e Tapentadol.
Description: Participants were requested to rate their tapentadol (new) analgesic medication on a 5-point scale. The medication was rated as excellent, very good, good, fair and poor.
Time Frame: After 6 weeks
Population: Intention to treat (ITT).
Measure: Number; unit: participants
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 55
participants
  Excellent | 3
  Very Good | 27
  Good | 21
  Fair | 4
  Poor | 0

18. Secondary Outcome: Participant's Satisfaction With New Analgesic Treatment, i.e Tapentadol.
Description: as for outcome 17
Time Frame: After 12 weeks
Population: Intention to treat (ITT).
Measure: Number; unit: participants
Arm/Group | Tapentadol PR
Number analyzed (Participants) | 32
participants
  Excellent | 3
  Very Good | 16
  Good | 12
  Fair | 1
  Poor | 0

19. Secondary Outcome: Mean Equipotency Ratio of Tapentadol Compared to Buprenorphine
Description: Tapentadol was compared to Transdermal Buprenorphine with Buprenorphine set to 1. The average total daily dose of Tapentadol at which a pain score equivalent or below to the pain score at the end of observation period under Transdermal Buprenorphine was reached was documented as the equipotent or equianalgesic dose to the total daily dose of the previously used Transdermal Buprenorphine.
Time Frame: Baseline; End of Week 6 (6 Weeks)
Population: Intention to treat (ITT). 48 participants with previous transdermal buprenorphine treatment.
Measure: Number; unit: Ratio
Groups:
- Tapentadol: All participants started with either 50 mg, 100 mg or 150 mg tapentadol hydrochloride PR (twice daily). The dose of tapentadol hydrochloride PR was adjusted to a level that provided adequate analgesia (upwards or downwards on a weekly basis as needed). After 5 weeks the doses of tapentadol hydrochloride PR was kept stable. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). Tapentadol hydrochloride IR 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes however, participants were not permitted to dose tapentadol hydrochloride IR once 500 mg tapentadol hydrochloride PR dose was reached.
Arm/Group | Tapentadol
Number analyzed (Participants) | 48
Ratio | 281.1

20. Secondary Outcome: Mean Equipotency Ratio of Tapentadol Compared to Oxycodone
Description: Tapentadol was compared to Oxycodone with Oxycodone set to 1. The average total daily dose of Tapentadol at which a pain score equivalent or below to the pain score at the end of observation period under Oxycodone was reached was documented as the equipotent or equianalgesic dose to the total daily dose of the previously used Oxycodone.
Time Frame: Baseline; End of Week 6 (6 Weeks)
Population: Intention to treat (ITT). 6 participants with previous oxycodone treatment.
Measure: Number; unit: Ratio
Arm/Group | Tapentadol
Number analyzed (Participants) | 6
Ratio | 4.6

ADVERSE EVENTS:
Time Frame: In total subjects were to be treated for up to 12 weeks with tapentadol.
Arm/Group | Tapentadol PR
Serious Adverse Events (participants affected / at risk) | 2/63
Other Adverse Events (participants affected / at risk) | 21/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol PR (N=63)
Abdominal pain (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Renal pain (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol PR (N=63)
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 8
Drug Withdrawal Syndrome (General disorders) | 4
Fatigue (General disorders) | 4
Dizziness (Nervous system disorders) | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Nausea (Gastrointestinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Grünenthal reserves the right to review any publication pertaining to the trial before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.